CLINICAL TRIAL: NCT07039136
Title: Feasibility and Usability of Immersive VR Mirror Therapy for Upper Limb Rehabilitation
Brief Title: Virtual Reality Mirrors Therapy Usability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assoc. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-FTR-RK-11
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Stroke
Keywords: Virtual Reality; Mirror Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Prospective parallel group with single-blinded design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Mirror Therapy Group (Experimental): Participants will receive virtual reality mirror therapy using head-mounted devices.
  Interventions: Other: Virtual Reality Mirror Therapy
- Sham Group (Sham Comparator): Participants will receive conventional mirror therapy with mirror box and then experience mirrored hand activities in virtual reality environment.
  Interventions: Other: Conventional Mirror Therapy; Other: Sham Virtual Reality

INTERVENTIONS:
Other: Virtual Reality Mirror Therapy — Participants will be seated on a chair with back support, their feet in contact with the ground, and both arms placed on a table. Data from participants' right forearms will be collected using Leap Motion tracking. In the virtual reality environment, both the original and mirrored forearms will be displayed within the participants' field of view.
  The mirror therapy session will consist of two 15-minute segments with a 10-minute rest period in between. Activities to be practiced during the session will include wrist flexion and extension, forearm pronation and supination, finger flexion and extension, finger opposition movements, squeezing a cloth, grasping a round object, wiping a table, and object manipulation. The therapy program will follow a progression from simple to complex and functional movements throughout the session. Session will begin with basic exercises such as flexion and extension movements of the fingers, wrist, and elbow, with 10 repetitions for each movement.
  Arms: Virtual Reality Mirror Therapy Group
Other: Conventional Mirror Therapy — Participants will be seated on a chair with back support, their feet in contact with the ground, and both arms placed on a table. Activities to be practiced during the session will include wrist flexion and extension, forearm pronation and supination, finger flexion and extension, finger opposition movements, squeezing a cloth, grasping a round object, wiping a table, and object manipulation. The therapy program will follow a progression from simple to complex and functional movements throughout the session. Session will begin with basic exercises such as flexion and extension movements of the fingers, wrist, and elbow, with 10 repetitions for each movement.
  Arms: Sham Group
Other: Sham Virtual Reality — Participants will experience virtual environments while seated and wearing a virtual reality headset, without interacting with the environment. The sham mirror therapy session will consist of two 15-minute segments with a 10-minute rest period in between.
  Arms: Sham Group

SUMMARY:
Mirror therapy has been shown to support motor recovery by stimulating neural mechanisms through visual feedback. Recent technological advancements, particularly in virtual reality (VR), have enabled the development of more immersive and interactive rehabilitation tools. This study focuses on evaluating the usability of a novel, Leap Motion-based Virtual Reality Mirror Therapy (VRMT) system designed to enhance upper limb rehabilitation in stroke patients by combining traditional mirror therapy principles with engaging, gamified digital environments.

DETAILED DESCRIPTION:
The VRMT system was developed to provide a low-cost, sensor-based rehabilitation tool that enables stroke survivors to engage in interactive upper limb exercises. Utilizing the Leap Motion sensor for real-time hand tracking, the system projects mirrored movements of the unaffected limb onto a virtual representation of the affected limb, reinforcing motor learning and neuroplasticity. The system includes multiple gamified tasks that simulate functional hand and arm movements within a virtual environment. Participants with subacute or chronic stroke used the system across several sessions, after which usability and user experience were assessed using standardized tools such as the System Usability Scale (SUS) and User Experience Questionnaire (UEQ). This approach allows for detailed feedback on comfort, satisfaction, interaction quality, and perceived effectiveness, contributing to future development and clinical integration of VR-based rehabilitation technologies.The aim of this study is to evaluate the usability, acceptability, and user experience of a Leap Motion-based Virtual Reality Mirror Therapy (VRMT) system designed to support upper limb rehabilitation in individuals with stroke. By integrating traditional mirror therapy principles with immersive virtual environments, the study seeks to determine the feasibility of using this system in clinical and home-based rehabilitation settings.

ELIGIBILITY:
Inclusion Criteria:

* Stereo acuity score of 3552 arc/sec in the Titmus Fly Test
* No prior virtual reality experience

Exclusion Criteria:

* Severe sensory impairments (vision or hearing)
* Being diagnosed with neurological disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Simulator Sickness Questionnaire | One hour
  "The SSQ evaluates 16 symptoms-including eye strain, nausea, sweating, and headache-using a four-point scale (none, mild, moderate, and severe). These symptoms are categorized into three overlapping subscales: nausea, oculomotor discomfort, and disorientation. Higher scores within each subscale reflect more intense experiences of simulator sickness. In military aviation contexts, a total SSQ score above 20 is typically interpreted as indicative of poor tolerance to simulation exposure. The total score generally ranges from 0 to 30, with higher scores indicating lower tolerance to simulated environments.

SECONDARY OUTCOMES:
Presence Questionnaire | One hour
  The PQ comprises four subscales: Involvement, Sensory Fidelity, Adaptation/Immersion, and Interface Quality. Participants respond to each item using a 5-phe total score generally ranges from 0 to 30, with higher scores indicating lower tolerance to simulated environments.oint Likert scale, reflecting their perceived experience in the virtual environment. The total score generally ranges from 24 to 168, with higher scores indicating better presence feeling in simulated environments.
Virtual Reality Sickness Questionnaire | One hour
  The PQ comprises four subscales: Involvement, Sensory Fidelity, Adaptation/Immersion, and Interface Quality. Participants respond to each item using a 5-phe total score generally ranges from 0 to 30, with higher scores indicating lower tolerance to simulated environments.oint Likert scale, reflecting their perceived experience in the virtual environment. The total score generally ranges from 0 to 27, with higher scores indicates higher motion sickness feeling in simulated environments.
System Usability Scale | One hour
  The System Usability Scale (SUS) is a 10-item instrument developed to rapidly assess the usability of various technological systems, including websites, software, hardware, and mobile devices. It employs a 5-point Likert scale and focuses primarily on user-perceived usability.A score of 68 is considered the average benchmark, with scores above this value indicating above-average usability, and scores below 68 reflecting below-average usability. Systems receiving the highest usability ratings fall into the A+ category, corresponding to the 96th to 100th percentile range.The total score generally ranges from 0 to 100, with higher scores indicates better usability..
Virtual Reality System Usability Questionnaire | One hour
  The Virtual Reality System Usability Questionnaire (VRSUQ), which has been previously applied in VR usability research, will be employed to assess system functionality and ease of interaction. The questionnaire includes items covering system control, interface design, and overall satisfaction. Responses are provided on a 5 point Likert-type scale ranging from strongly disagree to strongly agree. Higher scores reflect greater perceived usability and a more favorable user experience with the virtual environment .The total score generally ranges from 9 to 45

CONTACTS AND LOCATIONS:
Overall Officials: ramazan kurul, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (2):
- Turkey (Türkiye) (2):
  - Faculty of Health Sciences Bolu Abant Izzet Baysal University, Bolu, Merkez
  - Bolu Abant Izzet Baysal University Department of Physiotherapy and Rehabilitation, Bolu

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes will be shared.IPD will be available 6 months after publication of the main study results. Data will be shared with qualified researchers affiliated with academic or medical institutions, upon request and subject to ethical approval or data use agreements if applicable.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication, the study will be available indefinitely.
Access Criteria: Researchers may submit a data request by contacting the corresponding author via email. Approved users will receive access through a secure, password-protected institutional data-sharing platform or encrypted file transfer.